CLINICAL TRIAL: NCT02348983
Title: Weight Loss Intervention in Long-Haul Truck Drivers: A Pilot Study
Acronym: WHEEL-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Matthew Thiese, Assistant Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAP-ERC 5T42OH009229-06 Pilot
Record Dates: First submitted 2015-01-16; First posted 2015-01-28 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interventional Arm (Experimental): Health coaching arm to assess feasibility of intervention among truck driving population. Coaching will be weekly with emphasis on both diet and physical activity. No medication or treatment devices are administered.
  Interventions: Behavioral: Health Coaching via Telephone

INTERVENTIONS:
Behavioral: Health Coaching via Telephone — Health coaching arm to assess feasibility of intervention among truck driving population. Coaching will be weekly with emphasis on both diet and physical activity. No medication or treatment devices are administered.

SUMMARY:
Being obese can be a risk factor for many health problems, including high cholesterol, high blood pressure, low back pain, heart attacks and some cancers. Truckers, who are integral to our economy, face challenges that put them at increased likelihood of being obese. The investigators want to come up with a program to help drivers get to a healthy weight and stay there.

The WHEEL pilot study is a 12 week weight loss intervention in long-haul commercial truck drivers. The study involves two visits to the University of Utah's Rocky Mountain Center for Occupational and Environmental Health, one at the start of the study and a second one at the end of the study. Both visits include a general health history questionnaire, a 24-hour diet recall questionnaire, anthropometric measurements, as well as an assessment of blood pressure, hemoglobin A1c, and a cholesterol and lipid panel. Each truck driver is assigned a health coach who helps the driver create and achieve three health goals.

The health coach works with the driver to set individualized goals specific to weight loss, and contacts the driver weekly to check in and tweak goals as needed.

Drivers are also compensated for their participation in the study and get to keep all of the intervention materials that the investigators give them. All that the researchers ask is that they try their best to have a healthier lifestyle and give us feedback on what they liked and didn't like in the study.

DETAILED DESCRIPTION:
The investigators recruited 13 truckers based in Utah's Wasatch Front (population 2.2 Million) who expressed interest in participating in a weight loss intervention when they participated in the cross-sectional truck driver study (current enrollment, n= 817 truckers). Other options the investigators may pursue to maintain enrollment include enrolling participants directly through local trucking companies. Participants will be screened for eligibility based on

* Age > 21
* BMI > 30 kg/m2
* No reported unstable chronic disease

Interstate truckers are required to be at least 21 years old. Participants will not be enrolled in the intervention until they complete the physical assessment component of the baseline visit that includes blood pressure, lipids, and HbA1c. Individuals who do not meet the established medical guidelines and regulations of the FMCSA will be excluded. Those individuals will be advised to follow-up for care with their personal physicians, and/or will be referred to a primary care clinic.

Health coaches will have at least weekly contact with participants to discuss individual goals and behavior change. Motivational messages will be delivered in addition to weekly content via text messages and/or emails. Research suggests that individuals who begin losing weight quickly are more successful at weight loss and maintaining loss, therefore, after 3 weeks individuals who have not lost at least 3 pounds will receive additional contacts with health coaches to address slow rate of weight loss. Individual Competitions surrounding successful healthy behaviors of Truckers will be conducted every other week. Winning behaviors will be shared with other participants by email, text, phone calls, blogs and/or other distance friendly format to both engage drivers and model successful peer behaviors.

This is a study of weight loss intervention for long-haul commercial truck drivers who face unusual challenges to a healthy lifestyle while working. Participants (n=13) will be long-haul commercial truck drivers with a BMI over 30 kg/m2. Due to licensing issues, all interstate truck drivers are required to be at least 21 years old (US DOT, FMCSA), and thus proposed study participants will be at least 21 years old.

The investigators are aware that there are some intrastate truck drivers who may be under age 21, however they are a much smaller and different population. By definition they are not long-haul drivers, tend to have more job instability, have a different occupational environment that is relevant to this study (e.g., sleep at home), and thus are a different population that this research does not target. Thus, this study has sound rationale for not including children ages 18-20.

The sampling will be convenient. Participants will be recruited using email, postal mail and opportunities for personal contact that are identified through the Utah Trucking Association website, newsletter, at truck stops, and at Commercial Truck Driver meetings. The investigators will inquire for current interest among subjects from our current cross sectional study who indicated interest in a follow-up study.

Participants will be screened for approximate BMI, and medical history prior to recruitment. Participants under current treatment for cancer will be excluded. Participants with significant medical issues (such as unstable blood pressure, diabetes mellitus) will be asked to provide a medical release from their physician prior to participation. Participants currently in treatment for cancer will be excluded. In addition participants will not be enrolled until they have completed the physical assessment component of the study with blood pressure below 159/99 mm Hg (stage 2 hypertension), HbA1c below 10.0%, and total cholesterol below 300 mg/dL. If participants do not meet these standards a letter of permission to participate from a physician will be required. Participants will be referred to their personal physician or the primary care clinic at the University of Utah Redwood Health Center if they do not have a personal physician to obtain such permission.

Study visits will take place in the Occupational Medicine conference room at the University of Utah Redwood Health Center where Drs. Eric Wood practice, to gather demographic data, medical history, reported physical activity, occupational health outcomes (slips trips and falls) and psychosocial factors, self-efficacy, sleepiness scale, job satisfaction and measure blood lipids, hemoglobin A1c and HsCRP, and body weight and circumferences at baseline and 12 weeks for all participants t. Participants will weigh themselves weekly using a scale provided by the study and will report weekly weight to health coaches using a scale provided via telephone, text, or email. Participants will have at least weekly contact with research staff (health coaches) regarding the intervention in the first 12 weeks of WHEEL. Contact will continue bi-weekly after the first 12 weeks of WHEEL with a goal of continued weight loss or weight loss maintenance.

All participants will receive the weight loss intervention. Participants will be monitored closely for weight loss success in the first 3 weeks of the intervention. If weight loss is not at least 3 pounds, then health coaches will double their efforts with these participants as it is known that early success is associated with better long-term success.

The investigators will obtain information on questionnaires, asking a person's birth date, but only record a person's age in tenths of a year. The investigators will measure height, weight, waist, hip, chest, neck circumferences, blood pressure, heart rate, take a finger-stick to measure fasting glucose, hemoglobin A1c, highly sensitive C-Reactive Protein, and blood lipids using point of service analysis and perform a urinalysis. No blood specimens will be stored.

Measurements and questionnaires will be completed in the Occupational Medicine conference room at the University of Utah Redwood Health Center in Salt Lake City. This clinic is conveniently located around the corner from a large truck stop, and close to both I-80 and I-15, the two main interstates in Salt Lake City. The clinic has ample truck-friendly parking. The investigators have obtained letters of support from The Utah Trucking Association. Data will be recorded on laptop computers that are encrypted. Consent forms will be transported to the University of Utah for storage in locked cabinets.

ELIGIBILITY:
* Participants will be screened for eligibility based on:
* Age > 21
* BMI > 30 kg/m2
* No reported unstable chronic disease.
* Participants will not be enrolled in the intervention until they complete the physical assessment component of the baseline visit that includes blood pressure, lipids, and HbA1c.
* Individuals who do not meet the established medical guidelines and regulations of the FMCSA will be excluded. Those individuals will be advised to follow-up for care with their personal physicians, and/or will be referred to a primary care clinic.

Inclusion of women

Women will be included as they are represented in this population, although, the investigators expect, at rates that are less than the overall population. This is a convenience sample, thus there will not be attempts to over or under represent genders. The individualization of the interventions increases the likelihood of success of the intervention with both men and women.

Inclusion of minorities

The investigators will include minorities when possible. This is a convenience sample, so there will not be attempts to either over or under represent any racial or ethnic group.

Inclusion of Children

Commercial truck drivers must be 21 to drive interstate routes. Therefore, children, including those 18-20 years old, will not be included.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Measured Weight Loss from baseline to the end of the study | 12 weeks
  Difference in measured weight from baseline to the end of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Thiese MS, Effiong AC, Ott U, Passey DG, Arnold ZC, Ronna BB, Muthe PA, Wood EM, Murtaugh MA. A Clinical Trial on Weight Loss among Truck Drivers. Int J Occup Environ Med. 2015 Apr;6(2):104-12. doi: 10.15171/ijoem.2015.551. PMID 25890604